CLINICAL TRIAL: NCT03729739
Title: Comparison of Quantitative Flow Ratio (QFR) and Conventional Pressure-wire Based Functional Evaluation for Guiding Coronary Intervention. A Randomized Clinical Non-inferiority Trial
Brief Title: Functional Assessment by Virtual Online Reconstruction. The FAVOR III Europe Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Medis Medical Imaging Systems (Unknown)
Responsible Party: Principal Investigator, Evald Hoej Christiansen, Consultant cardiologist, Associate professor, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1-10-72-263-18
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Disease
Keywords: Fractional Flow Reserve (FFR); Quantitative Flow Ratio (QFR); Stable coronary artery disease; Angina pectoris; Angiography derived fractional flow reserve
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris

STUDY DESIGN:
Intervention Model Description: Randomized clinical non-inferiority trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QFR-based diagnostic strategy (Experimental): Intermediate stenosis with indication for evaluation are diagnosed by Quantitative flow ratio (QFR).
  Revascularization is indicated if QFR≤0.80. Treatment is performed according to standard clinical practice.
  Interventions: Diagnostic Test: QFR-based diagnostic strategy
- FFR-based diagnostic strategy (Active Comparator): Intermediate stenosis with indication for evaluation are diagnosed by fractional flow reserve (FFR).
  Revascularization is indicated if FFR≤0.80. Treatment is performed according to standard clinical practice.
  Interventions: Diagnostic Test: FFR-based diagnostic strategy

INTERVENTIONS:
Diagnostic Test: QFR-based diagnostic strategy — Novel computer based calculation of lesion severity. Pressure wire-free and adenosine-free
  Arms: QFR-based diagnostic strategy
Diagnostic Test: FFR-based diagnostic strategy — Standard FFR based diagnostic method. Pressure drop across the stenosis is measured with a pressure wire during medical induced hyperaemic conditions
  Arms: FFR-based diagnostic strategy

SUMMARY:
Quantitative Flow Ratio (QFR) is a novel method for evaluating the functional significance of coronary stenosis. QFR is estimated based on two angiographic projections. Studies have shown a good correlation with the present wire-based standard approach Fractional Flow Reserve (FFR) for assessment of intermediate coronary stenosis. The purpose of the FAVOR III Europe Japan study is to investigate if a QFR-based diagnostic strategy will results in non-inferior clinical outcome after 12 months compared to a standard pressure-wire guided strategy in evaluation of patients with chest pain (stable angina pectoris) and intermediate coronary stenosis.

DETAILED DESCRIPTION:
Patients at high risk of having one or more coronary stenosis are evaluated routinely by invasive coronary angiography (CAG). Lesions are often quantified by visual assessment of the angiogram, but physiological assessment of the functional significance by fractional flow reserve has been shown to improve clinical outcome, to reduce number of stents implanted, and has obtained the highest recommendation in European guidelines. FFR is assessed during CAG by advancing a wire with a pressure transducer towards the stenosis and measure the ratio in pressure between the two sides of the stenosis during medical induced maximum blood flow (hyperaemia).

The solid evidence for FFR evaluation of coronary stenosis and the relative simplicity in performing the measurements have supported adoption of an FFR based strategy but the need for interrogating the stenosis by a pressure wire, the small risks associated hereto, the cost of the wire, and the drug inducing hyperaemia has limited more widespread adoption.

Quantitative Flow Ratio is a novel method for evaluating the functional significance of coronary stenosis by calculation of the pressure drop in the vessel based on computation of two angiographic projections.

Two multi-center studies, the FAVOR II Europe-Japan and China studies evaluated the feasibility and diagnostic performance of in-procedure QFR, showing very good agreement between QFR and FFR.

The purpose of the FAVOR III Europe Japan study is to investigate if a QFR-based diagnostic strategy yields non-inferior 12-month clinical outcome compared to a standard pressure-wire guided strategy in evaluation of patients with stable angina pectoris and intermediate coronary stenosis.

Primary hypothesis: A QFR based diagnostic strategy results in non-inferior clinical outcome, assessed by a composite endpoint of all cause death, non-fatal myocardial infarction (MI) and unplanned revascularization after one year, compared to a strategy of pressure wire-based FFR for assessment of physiological significance of intermediate coronary artery stenosis.

Methods: Investigator initiated, 1:1 randomized, prospective, clinical outcome, non-inferiority, multi-center trial performed at up to 40 international sites with inclusion of 2000 patients.

Patients with stable angina pectoris or need for evaluation of non-culprit lesions after acute MI are enrolled. At least two angiographic projections are acquired during resting conditions. If the angiographic criteria are met, the patient is randomized to either a QFR- or an FFR-based diagnostic strategy.

Revascularization is performed according to best standard by percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG).

Patient follow-up is continued until 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years and above
* Both genders
* Indication for invasive coronary angiography
* Patients with stable angina pectoris, or assessment of secondary lesions in stabilized non-STEMI patients or assessment of secondary lesions in patients with prior STEMI and staged evaluation of secondary lesions.
* Able to provide written informed consent

Angiographic inclusion criteria

* Diameter stenosis of 40-90% diameter stenosis
* Vessel diameter of at least 2.5 mm and supplying viable myocardium
* Patients with restenosis in a native coronary artery can be included

Exclusion Criteria:

* Severely impaired renal function: Glomerular filtration rate (GFR) < 20 mL/min/1.73m²
* Life expectancy less than one year
* Cardiogenic shock or unstable haemodynamic state (Killip class III and IV)
* ST-elevation myocardial infarction (STEMI) within 24 hours
* Bypass graft to any target vessel
* Atrial fibrillation at the time of the procedure
* Chronic total occlusions of any vessel with possible or established indication for treatment
* Pregnancy or intention to become pregnant during the course of the trial
* Breast feeding
* Planned need for concomitant valvular or aortic surgery
* Left ventricular ejection fraction (LVEF) < 30%
* Previous inclusion in the FAVOR III trial
* Enrolled in another clinical study, and for this reason not treated according to present European Society of Cardiology guidelines, or the protocol treatment conflicts with the protocol treatment of FAVOR III
* Inability to tolerate contrast media
* Inability to tolerate Adenosine

Angiographic exclusion criteria

* Ostial right coronary artery > 50% diameter stenosis
* Left main coronary artery > 50% diameter stenosis
* Lesions properties indicative of myocardial bridging
* Bifurcation lesions with major (>1 mm) step down in reference size across the bifurcation
* Severe tortuosity of any target vessel
* Severe overlap in the stenosed segment
* Poor image quality precluding identification of vessel contours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2001 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient oriented composite endpoint (PoCE) | 12 months
  A composite endpoint of 1) all-cause mortality, 2) any myocardial infarction, and 3) any unplanned revascularization

SECONDARY OUTCOMES:
Target vessel failure | 1 month
  A composite of cardiac death, target vessel myocardial infarction and ischemic driven target vessel revascularization.
Target vessel failure | 12 months
  A composite of cardiac death, target vessel myocardial infarction and ischemic driven target vessel revascularization.
Target vessel failure | 24 months
  A composite of cardiac death, target vessel myocardial infarction and ischemic driven target vessel revascularization.
All-cause mortality | 1 month
  Total death includes cardiac death and other fatal categories such as cerebrovascular death, death from other cardiovascular disease (i.e. pulmonary embolism, dissection aortic aneurism will be included in this category), death from malignant disease, death from suicide, violence or accident, or death from other reasons.
All-cause mortality | 12 months
  Total death includes cardiac death and other fatal categories such as cerebrovascular death, death from other cardiovascular disease (i.e. pulmonary embolism, dissection aortic aneurism will be included in this category), death from malignant disease, death from suicide, violence or accident, or death from other reasons.
All-cause mortality | 24 months
  Total death includes cardiac death and other fatal categories such as cerebrovascular death, death from other cardiovascular disease (i.e. pulmonary embolism, dissection aortic aneurism will be included in this category), death from malignant disease, death from suicide, violence or accident, or death from other reasons.
Cardiac death | 1 month
  Encompasses death due to coronary heart disease including fatal myocardial infarction, sudden cardiac death including fatal arrhythmias and cardiac arrest without successful resuscitation, death from heart failure including cardiogenic shock, and death related the cardiac procedure within 28 days from the procedure. If death is not clearly attributable to other non-cardiac causes it is adjudicated as cardiac death
Cardiac death | 12 months
  Encompasses death due to coronary heart disease including fatal myocardial infarction, sudden cardiac death including fatal arrhythmias and cardiac arrest without successful resuscitation, death from heart failure including cardiogenic shock, and death related the cardiac procedure within 28 days from the procedure. If death is not clearly attributable to other non-cardiac causes it is adjudicated as cardiac death
Cardiac death | 24 months
  Encompasses death due to coronary heart disease including fatal myocardial infarction, sudden cardiac death including fatal arrhythmias and cardiac arrest without successful resuscitation, death from heart failure including cardiogenic shock, and death related the cardiac procedure within 28 days from the procedure. If death is not clearly attributable to other non-cardiac causes it is adjudicated as cardiac death
Myocardial infarction | 1 month
  Procedure and non-procedure related myocardial infarction. Protocol defined.
Myocardial infarction | 12 months
  Procedure and non-procedure related myocardial infarction. Protocol defined.
Myocardial infarction | 24 months
  Procedure and non-procedure related myocardial infarction. Protocol defined.
Target vessel myocardial infarction | 1 month
  As "any myocardial infarction", but with culprit lesion in index vessel.
Target vessel myocardial infarction | 12 months
  As "any myocardial infarction", but with culprit lesion in index vessel.
Target vessel myocardial infarction | 24 months
  As "any myocardial infarction", but with culprit lesion in index vessel.
Any unplanned revascularization | 1 month
  Coronary artery bypass grafting (CABG) or PCI of any lesion.
  Planned Revascularization:
  Revascularization is considered planned when it is decided at the time of the index procedure, based on the results of angiography and functional testing. Planned revascularization could be performed at the time of the index procedure or within 60 days. Such revascularization is considered as "primary" revascularization and is not considered as an endpoint. The "planned" status of the revascularization is adjudicated.
  Unplanned Revascularization:
  Revascularization is considered "unplanned" when not performed as part of standard care during the index procedure or if it is not planned as a staged procedure to occur within 60 days.
Any unplanned revascularization | 12 months
  Coronary artery bypass grafting (CABG) or PCI of any lesion.
  Planned Revascularization:
  Revascularization is considered planned when it is decided at the time of the index procedure, based on the results of angiography and functional testing. Planned revascularization could be performed at the time of the index procedure or within 60 days. Such revascularization is considered as "primary" revascularization and is not considered as an endpoint. The "planned" status of the revascularization is adjudicated.
  Unplanned Revascularization:
  Revascularization is considered "unplanned" when not performed as part of standard care during the index procedure or if it is not planned as a staged procedure to occur within 60 days.
Any unplanned revascularization | 24 months
  Coronary artery bypass grafting (CABG) or PCI of any lesion.
  Planned Revascularization:
  Revascularization is considered planned when it is decided at the time of the index procedure, based on the results of angiography and functional testing. Planned revascularization could be performed at the time of the index procedure or within 60 days. Such revascularization is considered as "primary" revascularization and is not considered as an endpoint. The "planned" status of the revascularization is adjudicated.
  Unplanned Revascularization:
  Revascularization is considered "unplanned" when not performed as part of standard care during the index procedure or if it is not planned as a staged procedure to occur within 60 days.
Any ischemia driven de novo revascularization | 1 month
  Coronary artery bypass grafting or PCI of a vessel that was not evaluated nor treated during the index procedure. In stable patients, ischemia should always be documented, using for example FFR, SPECT scan or MRI
Any ischemia driven de novo revascularization | 12 months
  Coronary artery bypass grafting or PCI of a vessel that was not evaluated nor treated during the index procedure. In stable patients, ischemia should always be documented, using for example FFR, SPECT scan or MRI
Any ischemia driven de novo revascularization | 24 months
  Coronary artery bypass grafting or PCI of a vessel that was not evaluated nor treated during the index procedure. In stable patients, ischemia should always be documented, using for example FFR, SPECT scan or MRI
Ischemia driven target vessel revascularization | 1 month
  Coronary artery bypass grafting (CABG) or PCI of a study vessel with documented ischemia. In stable patients, ischemia should always be documented, using for example FFR, SPECT scan or MRI
Ischemia driven target vessel revascularization | 12 months
  Coronary artery bypass grafting (CABG) or PCI of a study vessel with documented ischemia. In stable patients, ischemia should always be documented, using for example FFR, SPECT scan or MRI
Ischemia driven target vessel revascularization | 24 months
  Coronary artery bypass grafting (CABG) or PCI of a study vessel with documented ischemia. In stable patients, ischemia should always be documented, using for example FFR, SPECT scan or MRI
Ischemia driven treated target lesion revascularization | 1 month
  Coronary artery bypass grafting (CABG) or PCI of a study vessel with documented ischemia that was treated during index or planned staged procedure. In stable patients, ischemia should always be documented, using for example FFR, SPECT scan or MRI
Ischemia driven treated target lesion revascularization | 12 months
  Coronary artery bypass grafting (CABG) or PCI of a study vessel with documented ischemia that was treated during index or planned staged procedure. In stable patients, ischemia should always be documented, using for example FFR, SPECT scan or MRI
Ischemia driven treated target lesion revascularization | 24 months
  Coronary artery bypass grafting (CABG) or PCI of a study vessel with documented ischemia that was treated during index or planned staged procedure. In stable patients, ischemia should always be documented, using for example FFR, SPECT scan or MRI
Ischemia driven, measured segment revascularization | 1 month
  Coronary artery bypass grafting (CABG) or PCI of a study vessel that was evaluated by either FFR or QFR but not treated. In stable patients, ischemia should always be documented, using for example FFR, SPECT scan or MRI.
Ischemia driven, measured segment revascularization | 12 months
  Coronary artery bypass grafting (CABG) or PCI of a study vessel that was evaluated by either FFR or QFR (both treated and not treated). In stable patients, ischemia should always be documented, using for example FFR, SPECT scan or MRI.
Ischemia driven, measured segment revascularization | 24 months
  Coronary artery bypass grafting (CABG) or PCI of a study vessel that was evaluated by either FFR or QFR but not treated. In stable patients, ischemia should always be documented, using for example FFR, SPECT scan or MRI.
Ischemia driven measured segment de novo revascularization | 1 month
  Coronary artery bypass grafting (CABG) or PCI of a study vessel that was evaluated by either FFR or QFR but not treated. In stable patients, ischemia should always be documented, using for example FFR, SPECT scan or MRI.
Ischemia driven measured segment de novo revascularization | 12 months
  Coronary artery bypass grafting (CABG) or PCI of a study vessel that was evaluated by either FFR or QFR but not treated. In stable patients, ischemia should always be documented, using for example FFR, SPECT scan or MRI.
Ischemia driven measured segment de novo revascularization | 24 months
  Coronary artery bypass grafting (CABG) or PCI of a study vessel that was evaluated by either FFR or QFR but not treated. In stable patients, ischemia should always be documented, using for example FFR, SPECT scan or MRI.
Feasibility of QFR | 1 hour
  Percentage of successful QFR in patients allocated to a QFR based diagnostic strategy
Feasibility of FFR | 1 hour
  Percentage of successfully performed FFR measurements in vessels with attempted FFR (vessel level) Percentages of patients with successful FFR measurements (all attempted)
Number of lesion interrogated | 1 hour
  Total number of lesions diagnosed with either QFR or FFR during the procedure
Procedure time | 1 hour
  Time from introduction of the sheet until the sheet for coronary access is removed from the patient
Contrast volume | 1 hour
  Total volume of contrast used in the procedure
Fluoroscopy time | 1 hour
  Total fluoroscopy time for the procedure
Number of stents implanted | 1 hour
  Total number of stents implanted during the procedure. Stents implanted in a staged procedure are included

CONTACTS AND LOCATIONS:
Overall Officials: Evald H. Christiansen, Prof., Principal Investigator — Aarhus University Hospital, Denmark
Locations (35):
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus N
  - Gentofte Hospital, Hellerup
- France (7):
  - Institut Arnault Tzanck, Saint-Laurent-du-Var, Nice
  - GCS ES Axium - Parc Rambot, Aix-en-Provence
  - CHU de Lille, Lille University Hospital, Lille
  - Institut Cardiovasculaire Paris Sud (ICPS), Hopital Jacques Cartier, Massy
  - Hopital Haut-Leveque, Pessac, Pessac
  - Hôpital Privé Claude Galien, Quincy
  - Clinique Pasteur, Toulouse, Toulouse
- Germany (3):
  - Charite-Universitatsmedizin Berlin, Berlin
  - Elisabeth Krankenhaus, Essen
  - University Clinic Leipzig, Leipzig
- Italy (8):
  - Ospedale Maggiore, AUSL Bologna, Bologna
  - Azienda Ospedaliero-Universitaria di Ferrara, University of Ferrara, Ferrara
  - Azienda Ospedaliero Universitaria Federico II di Napoli, Naples
  - San Luigi Gonzaga University Hospital, Turin, Orbassano
  - Arcispedale S. Maria Nuova di Reggio Emilia, Reggio Emilia
  - Ospedale degli Infermi di Rimini, Rimini
  - Ospedale di Rivoli, Torino, Torino
  - Azienda Ospedaliera Universitaria integrata Verona, Verona
- Riga Stradini University Hospital, Riga, Latvia
- Hospital of Lithuanian University of Health Sciences Kauno Klinikos, Kaunas, Lithuania
- Netherlands (3):
  - VU University Medical Center, Amsterdam
  - Academic Medical Center (AMC), Amsterdam
  - HagaZiekenhuis, The Hague
- Medical University of Warsaw, Warsaw, Poland
- Spain (6):
  - Hospital Clinico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Clinico de Coruña, A Coruña
  - Hospital Lucus Agusti LUGO, Lugo
  - Hospital Clinico San Carlos, Madrid
  - Hospital Clinico Universitario de Valladolid, Valladolid
  - Hospital Álvaro Cunqueiro, Vigo
- Sahlgrenska University Hospital, Gothenburg, Sweden
- Barbera Stähli, Zurich, Zûrich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tu S, Westra J, Yang J, von Birgelen C, Ferrara A, Pellicano M, Nef H, Tebaldi M, Murasato Y, Lansky A, Barbato E, van der Heijden LC, Reiber JHC, Holm NR, Wijns W; FAVOR Pilot Trial Study Group. Diagnostic Accuracy of Fast Computational Approaches to Derive Fractional Flow Reserve From Diagnostic Coronary Angiography: The International Multicenter FAVOR Pilot Study. JACC Cardiovasc Interv. 2016 Oct 10;9(19):2024-2035. doi: 10.1016/j.jcin.2016.07.013. PMID 27712739
- [Background] Westra J, Andersen BK, Campo G, Matsuo H, Koltowski L, Eftekhari A, Liu T, Di Serafino L, Di Girolamo D, Escaned J, Nef H, Naber C, Barbierato M, Tu S, Neghabat O, Madsen M, Tebaldi M, Tanigaki T, Kochman J, Somi S, Esposito G, Mercone G, Mejia-Renteria H, Ronco F, Botker HE, Wijns W, Christiansen EH, Holm NR. Diagnostic Performance of In-Procedure Angiography-Derived Quantitative Flow Reserve Compared to Pressure-Derived Fractional Flow Reserve: The FAVOR II Europe-Japan Study. J Am Heart Assoc. 2018 Jul 6;7(14):e009603. doi: 10.1161/JAHA.118.009603. PMID 29980523
- [Background] Westra J, Tu S, Winther S, Nissen L, Vestergaard MB, Andersen BK, Holck EN, Fox Maule C, Johansen JK, Andreasen LN, Simonsen JK, Zhang Y, Kristensen SD, Maeng M, Kaltoft A, Terkelsen CJ, Krusell LR, Jakobsen L, Reiber JHC, Lassen JF, Bottcher M, Botker HE, Christiansen EH, Holm NR. Evaluation of Coronary Artery Stenosis by Quantitative Flow Ratio During Invasive Coronary Angiography: The WIFI II Study (Wire-Free Functional Imaging II). Circ Cardiovasc Imaging. 2018 Mar;11(3):e007107. doi: 10.1161/CIRCIMAGING.117.007107. PMID 29555835
- [Background] Xu B, Tu S, Qiao S, Qu X, Chen Y, Yang J, Guo L, Sun Z, Li Z, Tian F, Fang W, Chen J, Li W, Guan C, Holm NR, Wijns W, Hu S. Diagnostic Accuracy of Angiography-Based Quantitative Flow Ratio Measurements for Online Assessment of Coronary Stenosis. J Am Coll Cardiol. 2017 Dec 26;70(25):3077-3087. doi: 10.1016/j.jacc.2017.10.035. Epub 2017 Oct 31. PMID 29101020
- [Derived] Andersen BK, Sejr-Hansen M, Maillard L, Campo G, Ramunddal T, Stahli BE, Guiducci V, Serafino LD, Escaned J, Santos IA, Lopez-Palop R, Landmesser U, Dieu RS, Mejia-Renteria H, Koltowski L, Ziubryte G, Cetran L, Adjedj J, Abdelwahed YS, Liu T, Mogensen LJH, Eftekhari A, Westra J, Lenk K, Casella G, Van Belle E, Biscaglia S, Olsen NT, Knaapen P, Kochman J, Santos RC, Scarsini R, Christiansen EH, Holm NR. Quantitative flow ratio versus fractional flow reserve for coronary revascularisation guidance (FAVOR III Europe): a multicentre, randomised, non-inferiority trial. Lancet. 2024 Nov 9;404(10465):1835-1846. doi: 10.1016/S0140-6736(24)02175-5. Epub 2024 Oct 30. PMID 39488224